CLINICAL TRIAL: NCT01573325
Title: Health-Related Quality of Life in the Low Model for End-Stage Liver Disease (MELD) Pre Transplant Patient Candidate: A Pilot Study
Brief Title: HRQoL in the Low MELD Pre-tx Population
Acronym: LowMELD
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Loyola University (Other)
Responsible Party: Principal Investigator, Rebecca Duke, Transplant Surgery Nurse Practitioner, Northwestern University
Other Study IDs: STU00060397
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Cirrhosis of the Liver
Keywords: Cirrhosis of the liver; Pre-liver transplant Candidate; Depression; Poor social support; Liver disease symptoms; Health releated quality of life
MeSH Terms: conditions — Fibrosis; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe the HRQoL in those with MELD scores </= 15 in a single center for those who are pre-liver transplant candidates

DETAILED DESCRIPTION:
The liver organ allocation system was significantly revised in 2002, allowing a more objective prioritization of liver transplant candidates. The revised Model for End Stage Liver Disease (MELD) system is based primarily on laboratory test results. Candidates with MELD scores of less than 15 are considered to be low priority for cadaveric liver transplant and have limited treatment options. Yet patients with low MELD scores may suffer from an array of symptoms associated with liver disease such as fatigue, sleep disturbances, and depression - all of which erode health-related quality of life (HRQoL). No previous studies were found that examined HRQoL in low MELD transplant patients. A better understanding of the HRQoL of these patients will allow clinicians to better meet their needs. Therefore, the aims of the proposed pilot capstone project are to examine HRQoL and to identify demographic and clinical characteristics including liver-disease related symptoms, functional status, perceived social support, biological functioning and mental health associated with HRQoL in pre-liver transplant candidates with low MELD scores. The revised Wilson and Cleary Quality of Life Model will be used to guide the project. Fifty pre-transplant liver candidates with MELD scores < 15 will be enrolled in the descriptive, cross-sectional pilot study. Participants will complete a written questionnaire measuring perceived HRQoL and clinical characteristics. Descriptive and correlational statistics will be used to analyze the data. Findings from this project will identify trends in factors that contribute to a HRQoL of this population and provide the foundation for a larger future project.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a patient in the liver transplant clinic at Northwestern Memorial Hospital or one of its satellite clinics (including Washington, Illinois; Portage, Indiana; Glenview, Illinois, Oakbrook, Illinois; Joliet, Illinois)
2. Adult patient between the ages of 18-75
3. Ability to read and speak English
4. Must be a candidate for liver transplant per Northwestern Memorial Hospital liver transplant multidisciplinary committee
5. Model for End Stage Liver Disease (MELD) score ≤15
6. Cognitive ability to complete measures

Exclusion Criteria:

1. Non-English speaking
2. Those who have already received a liver transplant
3. Hepatic encephalopathy as evidenced by:

   1. Grade II or more West Haven Criteria or Adapted West Haven Criteria
   2. Evidence of Asterixis upon exam at time of consent (if consented in person)
4. Acute liver failure as etiology for liver disease.
5. MELD score > 15
6. Mental retardation or cognitive disabilities preventing completion of the written questionnaire

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who are a candidate for a liver transplant at Northwester Memorial Hospital with MELD score </=15
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Duke, MSN, Principal Investigator — Northwestern University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 Subjects were recruited from NMH clinic and satellite clinics. Recruitement was from 03/29/12 to 06/19/12
Groups:
- Study Popoulation: There was only one group as this was a descriptive prospective study. They all completed identical questionnaires including the Quality of Life Index, the Short-form Liver Disease Quality of Life tool, the Medical Outcomes Study Social Support Survey, the demographic tool and the Center for Epidemiological Studies Depression tool.
Period: Overall Study
Arm/Group | Study Popoulation
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Popoulation: There was only one group as this was a descriptive prospective study
Arm/Group | Study Popoulation
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.26 (10.774)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Perceived HRQoL Score. Overall Qualty of Life Index Tool Was Utilized.
Description: Describe perceived HRQoL in patients with low MELD scores (≤15) pre-liver transplant patient population. Overall Qualty of Life Index tool was utilized. The subscales were not utilized. The unit of measurement was scores on a scale. QLI tool has a range of 0-30 for total possible score. With the higher the score the higher the HRQoL.
Time Frame: 2-3 months
Population: Entire study population was analyzed
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Study Popoulation
Number analyzed (Participants) | 50
scores on a scale | 20.19 (5.98)

2. Secondary Outcome: Percentage of Subjects With Depressive Scores Who Had a Poor HRQoL
Description: Identify clinical characteristics such as environmental factors, patient biology, liver-disease related symptoms, functional status, general health perception, characteristics of the individual associated with perceived HRQoL in patients with low MELD scores (≤15) pre-transplant. What characteristics were found to be predictive of poor HRQoL. Tools utilized each assessed the specific variables including patient biology, liver disease symptoms, functional status, general health perception, and characteristics of the individual.
Time Frame: 2-3 months
Population: Entire study population was analyzed
Measure: Number; unit: percentage of participants
Arm/Group | Population Predicted by Have Poor HRQOL by Depressive Symptoms
Number analyzed (Participants) | 50
percentage of participants | 78

ADVERSE EVENTS:
Arm/Group | Study Popoulation
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

LIMITATIONS AND CAVEATS:
The small sample size and convenience sampling were limitations of this study. Additionally, since subjects were recruited from only one site, generalizability of findings is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No